CLINICAL TRIAL: NCT02523443
Title: A Prospective Randomized Controlled Clinical Trial of Patient Controlled Epidural Analgesia Versus Intravenous Patient Controlled Analgesia for Post-Operative Pain Control in Patients Undergoing Elective Open Liver Resection
Brief Title: Patient Controlled Epidural Analgesia Versus Intravenous Patient Controlled Analgesia for Post-Operative Pain Control in Patients Undergoing Elective Liver Resection
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-148
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Liver Cancer; Pain Management
Keywords: Epidural Analgesia; Intravenous Patient Controlled; 15-148
MeSH Terms: conditions — Liver Neoplasms; Agnosia | interventions — Analgesia, Patient-Controlled

ARMS (2):
- IV PCA after surgery (Active Comparator): general anesthesia with post-operative IV PCA with a standard demand pump
  Interventions: Other: IV PCA
- PCEA during and after surgery (Experimental): general anesthesia with post-operative thoracic epidural analgesia with a standard demand pump
  Interventions: Other: PCEA

INTERVENTIONS:
Other: IV PCA — Patients undergoing IV PCA for pain control will have intravenous (IV) analgesia provided through a demand pump started in the recovery room.
  Arms: IV PCA after surgery
Other: PCEA — Patients in this group will have the epidural catheter placed by the anesthesia pain service team in the pre-surgical center (PSC) as performed routinely at MSKCC. The epidural will be used intra-operatively at the end of liver resection phase of the surgical procedure, once the specimen has been extracted, and continued subsequently in the post-operative phase for pain management.
  Arms: PCEA during and after surgery

SUMMARY:
The purpose of this study is to learn whether patient-controlled epidural analgesia (PCEA) is a better method for managing pain after liver resection compared to patient-controlled analgesia (IV PCA). Currently, the standard pain control method for liver resection patients is IV PCA. There is not enough data on how epidural (PCEA) relieves pain and movement on a day to day basis after liver resection.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years or older) who are able to provide informed consent.
* Patients undergoing open elective liver resection for primary liver pathology (benign or malignant) or secondary metastatic liver disease, including patients undergoing concomitant surgical procedures (such as colorectal resection or debulking procedures), with no contraindication to the insertion of an epidural catheter (localized infection, septicemia, or pre-operative coagulopathy).

Exclusion Criteria:

* Patients with a history of documented anaphylaxis or contraindication to any of the study medications or standardized intra-operative medications. These include dilaudid, fentanyl, and bupivacaine.
* Patients with pain at rest or with movement measured by NRS >2.
* Patients receiving high dose opioids on a chronic basis (greater than or equivalent to 60mg of morphine per day).
* Patients with severe chronic obstructive pulmonary disease (COPD) defined as an FEV1 <50%.
* Patients with significant cognitive impairment or documented psychologic impairment.
* Contraindication to epidural catheter placement including bleeding diathesis (essential thrombocythemia, idiopathic thrombocytopenic purpura, von Willebrand disease, and hemophilia A or B), neurological dysfunction (multiple sclerosis, subacute myelo-opticoneuropathy or preexisting lower limb neurological deficit), prior extensive spinal surgery or major spinal deformity, pre-operative use of anti-coagulant with planned use of therapeutic dose of anti-coagulant in post-operatively, documented pre-operative coagulopathy (INR greater than 1.3 not on Coumadin or PTT greater than 42), platelets less than 100,000/μL, or evidence of infection at potential epidural site.
* Cirrhotic patients. When incidentally discovered intra-operatively, patients will be excluded from the study and replaced, but will be followed for primary and secondary endpoints.
* Patients with poor performance status preoperatively such that they are unable to walk up two flights of stairs.
* Patients taking any opioid agonist/antagonist medication (i.e. Buprenorphine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
ability to detect a 2-point NRS scale difference | 1 year
  The primary endpoint assesses differences in pain control between PCEA and IV PCA after a "get up and go" test performed on POD2 during pain rounds, evaluated using a NRS pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Vittoria Arslan-Carlon, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/